CLINICAL TRIAL: NCT07288086
Title: Reliability and Effectiveness of New Enova Preloaded Intaocular Lens and Cartridge System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Semih Çakmak, Assistant Professor, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulUni
Record Dates: First submitted 2025-08-26; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cataract Surgery; Intraocular Lens
Keywords: cataract surgery; intraocular lens; preloaded intraocular lens; Enova

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who need cataract surgery (Experimental): Participants will undergo standard cataract surgery using the new preloaded intraocular lens (IOL) system. The intervention involves implantation of the preloaded IOL following routine phacoemulsification techniques.
  Interventions: Device: Preloaded intraocular lens system

INTERVENTIONS:
Device: Preloaded intraocular lens system — This intervention uses a preloaded IOL delivery system, which allows for a single-use, sterile implantation during standard phacoemulsification cataract surgery. Unlike standard manually loaded IOLs, this system reduces preparation time and minimizes handling of the lens, potentially improving surgical efficiency and maintaining lens sterility.

SUMMARY:
Evaluation of the safety and efficacy of the new Enova® preloaded monofocal intraocular lens and cartridge injector system in cataract surgery

DETAILED DESCRIPTION:
In this prospective and single-center clinical study, the safety and efficacy of the Enova PGF3 intraocular lens (IOL) and cartridge injector system will be evaluated.

The Enova PGF3 cartridge injector system is designed to be used in cataract surgeries. Cataract patients aged 40 years and older, both male and female, without any serious ocular disease other than cataracts, will undergo IOL implantation following cataract surgery. It is planned to perform a total of 200 implantations with either unilateral or bilateral implantation of the participants' eyes.

Postoperative visual acuity, refraction, patient satisfaction, and adverse events will be monitored during follow-up visits at day 1, week 1, and month 1.

The primary objectives of the study are to achieve an uncorrected distance visual acuity of 20/20 or better, and to maintain an error and complication rate related to the preloaded system below 7.5%. Secondary objectives include evaluating patient satisfaction and assessing whether surgeons find the preloaded system easy to use and if it meets their expectations.

The primary endpoints are refractive stability within ±0.50 D, uncorrected distance visual acuity of 20/20 or better, and a general clinical performance rating of the preloaded system with a score of 95% or higher. Secondary endpoints include the duration of surgery, accuracy of lens positioning, surgical complications, surgeon-reported ease of use, and patient satisfaction survey results meeting expectations.

As a safety parameter, adverse events reported in postoperative surgical reports will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adults of either sex.

Age 40 years or older.

Willing and able to provide written informed consent and comply with planned study visits and procedures.

Healthy ocular status, with no ocular pathology other than cataract and mild refractive error.

Potential visual acuity of 20/32 (0.2 logMAR) or better in both eyes.

Presence of regular corneal astigmatism suitable for treatment with the study device.

Candidates for uncomplicated cataract surgery using the study device.

Exclusion Criteria:

* Irregular corneal astigmatism (e.g., keratoconus).

Corneal pathology (e.g., scar, dystrophy, pterygium, moderate to severe dry eye).

Monocular conditions (e.g., amblyopia).

Previous corneal surgery, including radial keratotomy, corneal refractive surgery, corneal transplantation, DSAEK, or lamellar keratoplasty.

Previous anterior or posterior segment surgery (e.g., vitrectomy, laser iridotomy).

Diabetic retinopathy.

Macular pathology (e.g., age-related macular degeneration [ARMD], epiretinal membrane [ERM]).

History of retinal detachment.

Surgical complications that may affect study outcomes, such as:

Decentration due to capsulorhexis issues

Improper lens placement

Inadequate or missing postoperative capsular support

Posterior capsular rupture

Vitreous loss

Iris damage (tear, rupture, etc.)

Acute or chronic ocular diseases known to affect visual acuity or study outcomes (e.g., immunosuppressed state, connective tissue disease, clinically significant atopic disease, diabetes, or other systemic or ocular conditions).

Participation in any investigational drug or device study within 30 days prior to study start, or ongoing participation in another study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Distance Visual Acuity (UDVA) - Photopic Conditions | 1 month postoperatively
  Proportion of eyes achieving 20/20 or better uncorrected distance visual acuity under photopic conditions.
Subjective Refractive Error | 1 month postoperatively
  Eyes with a postoperative refractive error within ±0.50 diopters of the intended target.
Overall Clinical Performance of the Preloaded IOL System | 1 month after surgery
  Surgeon-rated assessment of the general clinical performance of the preloaded system by The ENOVA PGF3 Questionnaire. This questionnaire is a 14-item, study-specific, non-validated survey developed to evaluate surgeons' experience with an intraocular lens (IOL) preloaded delivery system. Eleven items are rated on a 5-point Likert scale with the following scoring structure:
  1. = Low
  2. = Below Expectation
  3. = Meets Expectation
  4. = Above Expectation
  5. = Outstanding Performance
  Some additional items are Yes/No questions and do not contribute to the numerical total score.
  The total numerical score is calculated by summing the 11 Likert-scaled items. Total score range: 11 to 55, with higher scores indicating better performance and more favorable user experience.

SECONDARY OUTCOMES:
Preloaded System Evaluation Patient Questionnaire | Baseline (preoperative) and 1 month postoperatively
  Patient-reported outcomes assessing whether expectations for visual improvement and overall satisfaction were met.The questionnaire consists of 14 items assessing a patient's self-reported difficulty in performing vision-related daily activities. Each activity is rated using a 0-4 scale, where:
  4 = No difficulty
  3 = Mild difficulty
  2 = Moderate difficulty
  1 = Severe difficulty
  0 = Unable to perform the activity
  The total score is calculated by summing responses across all 14 items. Total possible score range: 0 to 56
  Higher scores indicate better visual function and less activity limitation.
  Lower scores indicate worse visual function.
Surgical Procedure Assessment | Intraoperative
  Surgeon-reported ease of lens implantation and accuracy of lens placement, evaluating whether expectations for procedural handling were met.The surgeon notes, during the operative visit, the location of the incision, the size of the incision, whether the implantation system is compatible with the wound site, how many seconds the implantation time is shortened, and whether there were any issues with the unfolding of the intraocular lens or its placement into the capsular bag.

OTHER OUTCOMES:
Serious Adverse Events | 1 month postoperatively
  Any serious adverse events occurring during surgery or within 1 month after surgery.
Postoperative Inflammation | 1 week and 1 month postoperatively
  Assessment of inflammation levels by biomicroscopic anterior chamber and vitreus examination according to Standardization of Uveitis Nomenclature (SUN) International Workshop Grading System
Intraocular Pressure, | 1 week and 1 month postoperatively
  Intraocular pressure is assessed via Goldmann Applanation Tonometry. Normal levels are accepted as 10-21 mmHG.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Istanbul Medical Faculty Ophthalmology Department, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared outside the study.

REFERENCES:
- [Result] Oshika T, Wolfe P. In vitro comparison of delivery performance of 4 preloaded intraocular lens injector systems for corneal and sclerocorneal incisions. J Cataract Refract Surg. 2019 Jun;45(6):840-846. doi: 10.1016/j.jcrs.2018.10.050. Epub 2019 Mar 8. PMID 30853318
- [Result] Joshi RS. Comparative evaluation of an automated preloaded delivery system with a non-preloaded system. Indian J Ophthalmol. 2022 Dec;70(12):4307-4311. doi: 10.4103/ijo.IJO_1635_22. PMID 36453335
- [Result] Acar B, Torun IM, Acar S. Evaluation of Preloaded IOL Delivery System and Hydrophobic Acrylic Intraocular Lens in Cataract Surgery. Open Ophthalmol J. 2018 Jun 14;12:94-103. doi: 10.2174/1874364101812010094. eCollection 2018. PMID 30008971